CLINICAL TRIAL: NCT04869293
Title: Assessment of Analgesia Through Hypnosis With 3D Virtual Reality During Extra-corporeal Lithotripsy (LAHMA)
Brief Title: Lithotripsy and Analgesia With 3D Hypnosis Mask
Acronym: LAHMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: GAMIDA (Unknown); Healthy Mind (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200879; IDRCB 2020-A02052-37 (Other: ANSM)
Record Dates: First submitted 2021-03-19; First posted 2021-05-03 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Renal Calculi; Pain
Keywords: therapeutic virtual reality; hypnosis
MeSH Terms: conditions — Kidney Calculi; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D virtual reality (Experimental): Use of Hypnosis 3D virtual reality headset
  Interventions: Device: Hypnosis 3D virtual reality headset
- Control (No Intervention): Standard of care : no hypnosis 3D virtual reality headset but a noise cancelling headphone

INTERVENTIONS:
Device: Hypnosis 3D virtual reality headset — 3D experience to journey through a natural and therapeutic environment. Immersion is amplified by the realism of 3D environment, a soothing sound atmosphere and specific medical hypnosis.
  Arms: 3D virtual reality

SUMMARY:
The study is a randomised trial of hypnosis with 3D virtual reality headset (intervention group) versus control group with no hypnosis and no virtual reality headset to compare remifentanil consumption during shock wave lithotripsy.

DETAILED DESCRIPTION:
The study is for patients undergoing shock wave lithotripsy in outpatient surgery unit.

It is proposed that using hypnosis with 3D virtual reality headset will reduce the requirements for intravenous remifentanil in a randomised controlled trial of one hundred and six patients.

Remifentanil is an opioid commonly used for lithotripsy. Shock wave lithotripsy is a commonly performed procedure associated with moderate pain and anxiety, in outpatient surgery unit. Opioids can cause unfavourable side-effects, most notably respiratory depression, sedation, nausea and vomiting

It is expected that by using 3D virtual reality to reduce pain and anxiety, there will be a reduced requirement for intravenous remifentanil.

The study will measure the dose of remifentanil required by patients randomised to receive either hypnosis with 3D virtual reality headset (intervention) or no hypnosis and no 3D virtual reality headset (control group).

Patients will be followed up prior to hospital discharge to assess their remifentanil use and pain, anxiety, comfort and their satisfaction with 3D virtual reality headset.

This new device is a non-pharmacological adjunct and can reduce pain intensity during procedure, reduce opioid use and length of stay in hospital and improve the patient experience whilst potentially reducing complications of intravenous opioid.

This study findings will be of interest for patients involved in surgery or investigative procedures normally carried out with intravenous opioids or sedation.

ELIGIBILITY:
Inclusion Criteria:

- Shock wave lithotripsy and outpatient surgery

Exclusion Criteria:

* Epilepsy
* Deafness, Blindness
* Schizophrenia, Hallucinations
* No french-speaking
* Autistic
* Motion sickness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Remifentanil use | Hour 1
  Remifentanil consumption (microgram) during shock wave lithotripsy

SECONDARY OUTCOMES:
Maximal level of pain during shock wave lithotripsy | Hour 1
  Use of analogical visual pain self-assessment at the end of the shock wave lithotripsy

CONTACTS AND LOCATIONS:
Overall Officials: Darless Clausse, MD, Principal Investigator — Hôpital européen Geroges-Pompidou
Locations (2):
- France (2):
  - Assistance Publique Hôpitaux de Paris, Necker, Paris
  - Assistance Publique Hôpitaux de Paris, Hôpital Européen Georges Pompidou, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team. Collaboration will be fostered.
  Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Eijlers R, Utens EMWJ, Staals LM, de Nijs PFA, Berghmans JM, Wijnen RMH, Hillegers MHJ, Dierckx B, Legerstee JS. Systematic Review and Meta-analysis of Virtual Reality in Pediatrics: Effects on Pain and Anxiety. Anesth Analg. 2019 Nov;129(5):1344-1353. doi: 10.1213/ANE.0000000000004165. PMID 31136330
- [Background] Scapin S, Echevarria-Guanilo ME, Boeira Fuculo Junior PR, Goncalves N, Rocha PK, Coimbra R. Virtual Reality in the treatment of burn patients: A systematic review. Burns. 2018 Sep;44(6):1403-1416. doi: 10.1016/j.burns.2017.11.002. Epub 2018 Feb 1. PMID 29395400
- [Background] Chan E, Foster S, Sambell R, Leong P. Clinical efficacy of virtual reality for acute procedural pain management: A systematic review and meta-analysis. PLoS One. 2018 Jul 27;13(7):e0200987. doi: 10.1371/journal.pone.0200987. eCollection 2018. PMID 30052655